CLINICAL TRIAL: NCT04620941
Title: Use of Reticulocyte Ratio and Neutrophil / Lymphocyte Ratio in the Diagnosis of Ventilator-associated Pneumonia
Status: Completed | Type: Observational
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Eylem Yaşar, Muğla Sıtkı Koçman University Department of Anesthesiology Specialist, Muğla Sıtkı Koçman University
Other Study IDs: 27/12/2019-19/XI
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Ventilator-associated Pneumonia (VAP)
Keywords: Ventilator-associated pneumonia; reticulocyte/hemoglobin ratio; neutrophil/lymphocyte ratio
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Reticulocyte Count

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ventilator-associated pneumonia: Ret-He values will be studied on the day (1st day), 4th and 7th days of VID diagnosis in patients receiving mechanical ventilation support in the intensive care unit. The hemogram, CRP, and NLR values that are routinely studied in the intensive care unit will be recorded. In addition, in case of infection, the routinely studied procalcitonin value will also be recorded. The patient's age, gender, APACHE II, SOFA scores will be recorded; respiratory system examination, fever, the mental status evaluation will be done daily.
  Interventions: Diagnostic Test: reticulocyte/hemoglobin (Ret-He) ratio

INTERVENTIONS:
Diagnostic Test: reticulocyte/hemoglobin (Ret-He) ratio — Ret-He values will be studied on the day (1st day), 4th and 7th days of the diagnosis of ventilator-associated pneumonia in patients hospitalized in the intensive care unit.

SUMMARY:
In this study, the utility of changes in the ratio of Ret-He and NLR as an early inflammation marker for VAP will be evaluated.

DETAILED DESCRIPTION:
Ventilator-associated pneumonia (VAP) is one of the most common nosocomial infections in the intensive care unit, affecting one third of patients requiring mechanical ventilation for a noninfectious reason. In the case of inflammation, iron retention increases in the reticuloendothelial system cells; hemoglobin (Hb) synthesis is reduced. It has been reported that the ratio of reticulocyte / hemoglobin (Ret-He) decreases in the early period in community-acquired pneumonia patients and may be a guide as a marker of inflammation. In addition, the neutrophil / lymphocyte ratio (NLR) is a parameter studied in the hemogram panel. It provides a clue to both the presence of infection and the focus of the infection.

In this study, the utility of changes in the ratio of Ret-He and NLR as an early inflammation marker for VAP will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

-Patients who need mechanical ventilation for longer than 48 hours for a noninfectious reason in the intensive care unit

Exclusion Criteria:

* Pulmonary or extrapulmonary infection before mechanical ventilation,
* severe immunosuppression,
* bleeding in the gastrointestinal system,
* using corticosteroids,
* neoplastic disease history

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who need mechanical ventilation for longer than 48 hours for a noninfectious reason in the intensive care unit
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Early inflammation markers for VAP | 7 days
  To investigate the use of NLR and Ret-He value as early inflammation markers for VAP.

SECONDARY OUTCOMES:
morbidity and mortality | 7 days
  To compare the effects of Ret-He and NLR values on morbidity and mortality with other inflammation markers

CONTACTS AND LOCATIONS:
Overall Officials: turhan togan, Study Chair — Mugla Sitki Kocman Universty Department of Infection Disease; Canan Gursoy, Study Chair — Mugla Sitki Kocma University Department of Intensive Care; Semra Demirbilek, Study Chair — Mugla Sitki Kocman Universty Department of Anesthesia
Locations (1):
- Mugla Sitki Kocman Universty, Muğla, Kötekli, Turkey (Türkiye)